CLINICAL TRIAL: NCT03117192
Title: Zinc Supplementation on Cellular Immunity in Thalassemia Major
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 02
Record Dates: First submitted 2017-03-31; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Thalassemia; Splenectomy; Status; Immunosuppression
Keywords: zinc supplementation; immunity; thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: This interventional study is a randomized controlled trial comparing the parallel provision of zinc and placebo in 2 groups of splenectomized thalassemia major patients.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Secretary to the department held an envelope that shows sample allocation after randomization. The envelope is only revealed after data gathering is finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc sulfate (Experimental): Zinc sulfate is provided in the form of syrup at a dose of 1.5 mg/kg/day, maximum 50 mg/day.
  Interventions: Drug: Zinc Sulfate
- Sucrose syrup (Placebo Comparator): Sucrose syrup is used as placebo, its provided in the form of syrup with similar appearance and taste.
  Interventions: Drug: Sucrose Syrup

INTERVENTIONS:
Drug: Zinc Sulfate — Zinc supplementation in syrup form
  Arms: Zinc sulfate
Drug: Sucrose Syrup — Sucrose as placebo, with same taste and consistency as zinc
  Arms: Sucrose syrup

SUMMARY:
Randomized controlled trial was conducted in post-splenectomy patients aged >12 years. Subjects are randomly assigned to two groups (zinc and placebo). 1.5 mg/kg/day (max 50 mg/day) of Zinc is administered.

DETAILED DESCRIPTION:
Thalassemia refers to a hereditary anaemic condition that occurs due to a single gene disorder resulting in a defect in globin production. Infection is an important cause of morbidity and mortality among thalassemia patients worldwide. Thalassemia patients are more prone to infection. Mechanism of this susceptibility is related to altered immune response compounded by splenectomy procedures common in patients with thalassemia. Zinc on the other hand plays important role in immune responses. This study aims to identify zinc supplementation to cellular immunity of splenectomized patients.

Randomized controlled trial was conducted in post-splenectomy patients aged >12 years. Subjects are randomly assigned to two groups (zinc and placebo). 1.5 mg/kg/day (max 50 mg/day) of Zinc is administered. Anamnesis, physical examination, and laboratory results such as peripheral blood, ferritin, transferrin saturation, serum zinc, immunologic markers for cellular immunity (lymphocyte count, CD4+ and CD8+ T lymphocyte count and functions) are evaluated at the start and end of the 12-week study.

Improvement in immune response is defined as an increase in the T lymphocyte count and CD4+ T lymphocyte count, decrease in CD8+, and increase in the CD4+/CD8+ ratio.12 The mean reference value for CD4+/CD8+ ratio is 1.4 (SD 0.6).15 CD4+ T lymphocyte function refers to its ability to synthesize IL-2 and TNF-α following exposure to 100 µL phytohaemagglutinin with proportions measured using flow cytometry. Meanwhile, CD8+ T lymphocyte function refers to its ability to synthesize IL-2 and TNF-α following exposure to 100 µL phytohaemagglutinin measured using flow cytometry.

The frequency of blood transfusion is calculated from the medical records of the subjects during the past 1 year, which is grouped as follows:

1. Seldom receive blood transfusions, if within a time period of one year the subject received blood transfusions of < 1 time.
2. Sometimes receive blood transfusions, if within a time period of one year the subject received blood transfusions of 2 - 3 times.
3. Often receive blood transfusions, if within a time period of one year the subject received blood transfusions of > 4 times.

Analysis was conducted using Statistical Package for Social Sciences (SPSS) version 20.0. Changes in immunologic parameters between the two groups that are numeric will be analysed using paired t-test for variables with a normal distribution, and Mann-Whitney test for numeric variables with non-normal distributions.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia major patients
* Age > 12 years
* Agreed to participate and signed the informed consent
* No other comorbidity beside thalassemia

Exclusion Criteria:

* HIV positive patients
* Those in steroid medication

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

PRIMARY OUTCOMES:
Patient's T-lymphocyte count | 12 weeks
  Measurement of patients CD4+ and CD8+ T-lymphocyte count in uL

CONTACTS AND LOCATIONS:
Overall Officials: Teny T Sari, M.D., PhD, Principal Investigator — Faculty of Medicine University of Indonesia
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No